CLINICAL TRIAL: NCT06371378
Title: Evaluation of the Effect of Different Peep Values on Gastric Residual Volume and Pulmonary Aspiration Risk in Patients Undergoing Spinal Surgery in Prone Position
Brief Title: Effect of Different Peep Values on Gastric Residual Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Süleyman Taygurt, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: gastric residual volume
Record Dates: First submitted 2024-02-01; First posted 2024-04-17 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Aspiration of Gastric Content
Keywords: prone position; Gastric POCUS (Point of Care Ultrasound); antrum diameter; risk of pulmonary aspiration; different peep levels

STUDY DESIGN:
Intervention Model Description: We gave three different peep values on the mechanic ventilator; 3 groups: Group I: PEEP O, Group II: PEEP 4, Group III: PEEP 8
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP I: PEEP 0 (Active Comparator): Patients will receive 0 cmH20 PEEP
  Interventions: Procedure: PEEP 0
- GROUP II: PEEP 4 (Active Comparator): Patients will receive 4 cmH20 PEEP
  Interventions: Procedure: PEEP 4
- GROUP III: PEEP 8 (Active Comparator): Patients will receive 8 cmH20 PEEP
  Interventions: Procedure: PEEP 8

INTERVENTIONS:
Procedure: PEEP 0 — PEEP 0 CMH20 will be used During Surgery
  Other Names: antrum diamater radio , gastric reziduel volume
  Arms: GROUP I: PEEP 0
Procedure: PEEP 4 — PEEP 4 CMH20 will be used During Surgery
  Arms: GROUP II: PEEP 4
Procedure: PEEP 8 — PEEP 8 CMH20 will be used During Surgery
  Arms: GROUP III: PEEP 8

SUMMARY:
The aim of this study was to predict the effect of gastric antrum diameter before extubation on intra-abdominal pressure changes and consequently on the risk of pulmonary aspiration in patients undergoing elective spinal surgery under general anaesthesia in the prone position in the Neurosurgery Operating Theatre of the Ministry of Health Ankara City Hospital and to take precautions accordingly. Gastric antrum diameter and intraabdominal pressure measurements may contribute to the improvement of anaesthetic practice by reducing the risk of pulmonary aspiration and additional complications.

DETAILED DESCRIPTION:
Prone positioning in spinal surgery is a very important issue for anaesthetists. Although there are many conditions that are taken into consideration in patient follow-up, it is a position frequently used in the treatment of pulmonary diseases other than surgery. PEEP application in the prone position is especially used in the treatment of conditions such as acute respiratory distress syndrome (ARDS). This treatment method basically aims to improve oxygenation and ventilation in the lungs. While providing improvement in the lungs, it may indirectly lead to some changes in the gastrointestinal system. Depending on PEEP levels, intra-abdominal pressure may increase and subsequently cause reflux of gastric contents or gastroparesis. The prone position itself also increases the risk of reflux. Gastric POCUS (Point of Care Ultrasound) is a noninvasive method that gives us information about the stomach contents and can be easily performed at the bedside. Both patient position and respiratory parameters, such as PEEP, may have an effect on gastric POCUS. Visualization of gastric content or detection of gastric retention allows us to predict possible pulmonary aspiration complications before extubation, and gastric POCUS may be a valuable marker before extubation in patients who remain in prone positions for a long time. The aim of this study was to determine the effect of PEEP application on the antrum diameter evaluated by gastric POCUS and the risk of aspiration before extubation in patients undergoing spinal surgery in the prone position.

ELIGIBILITY:
Inclusion Criteria

* 18-65 years of age
* ASA I-II risk group

Exclusion Criteria:

* Asthma
* COPD
* Gastroesophageal reflux
* Gastric herniation
* Gastric surgery,
* Intracranial tumor
* Epilepsy
* Neuromuscular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Gastric antrum diameter | induction of anaesthesia at 0 minutes,After induction of anaesthesia at 1 minutes,at 10 minutes at the end of the case
  Cross-sectional area (CSA) (cm2)

SECONDARY OUTCOMES:
Intraabdominal pressure (IAP) measurement | induction of anaesthesia at 0 minutes,After induction of anaesthesia at 1 minutes,at 10 minutes at the end of the case
  Comparing IAP between three groups.
gastric volume measurement | induction of anaesthesia at 0 minutes,After induction of anaesthesia at 1 minutes,at 10 minutes at the end of the case
  gastric volume (ml)

OTHER OUTCOMES:
Vital parameters Pulse oximetry (%) | induction of anaesthesia at 0 minutes,After induction of anaesthesia at 1 minutes,at 10 minutes at the end of the case
  Pulse oximetry (%)
Vital parameters systolic and diastolic blood pressure (mmHg) | induction of anaesthesia at 0 minutes,After induction of anaesthesia at 1 minutes,at 10 minutes at the end of the case
  systolic and diastolic blood pressure (mmHg)
Vital parameters heart rate (beats/minute) | induction of anaesthesia at 0 minutes,After induction of anaesthesia at 1 minutes,at 10 minutes at the end of the case
  heart rate (beats/minute)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chui J, Craen RA. An update on the prone position: Continuing Professional Development. Can J Anaesth. 2016 Jun;63(6):737-67. doi: 10.1007/s12630-016-0634-x. Epub 2016 Apr 12. PMID 27072147
- [Background] Fujishima S. Guideline-based management of acute respiratory failure and acute respiratory distress syndrome. J Intensive Care. 2023 Mar 10;11(1):10. doi: 10.1186/s40560-023-00658-3. PMID 36895001
- [Background] El-Boghdadly K, Wojcikiewicz T, Perlas A. Perioperative point-of-care gastric ultrasound. BJA Educ. 2019 Jul;19(7):219-226. doi: 10.1016/j.bjae.2019.03.003. Epub 2019 Apr 24. No abstract available. PMID 33456894